CLINICAL TRIAL: NCT06963099
Title: Use of Intra-corneal Ring Segments in Management of Non-ectatic Corneas With High Cylinder
Brief Title: INTACS for Non Ectatic With High Cylinder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elshimaa A.Mateen (Other)
Responsible Party: Sponsor-Investigator, Elshimaa A.Mateen, Assistant Professor, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-4-2PD
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High cylinder group (Other)
  Interventions: Other: INTACS implantation

INTERVENTIONS:
Other: INTACS implantation — intra corneal segments implantation

SUMMARY:
Intra-corneal rings implantation for correcting high cylinder errors in non ectatic corneas

ELIGIBILITY:
Inclusion Criteria:

* Non ectatic corneas with high cylinder error

Exclusion Criteria:

* Corneal ectasia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change of (1)visual acuity in log mar (2) keratometry readings in diopter 1) refraction. 2)High order aberrations | six months
  Using: (1) auto-refractometer (2) pentacam to assess keratometry changes.
changes of corneal parameters (K1.K2,K max) in diopter | six months
  Comparing pentacam readings pre and post operative.

CONTACTS AND LOCATIONS:
Locations (1):
- Elshimaa A.Mateen, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No